CLINICAL TRIAL: NCT06493422
Title: Online Interplay Between Deciding and Acting With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Joshua Cashaback, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2026374-5; U54GM104941 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-07-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Reaching; Brain; Decisions
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reaching task (Experimental): Mild cognitive impairment participants will make decisions while moving
  Interventions: Behavioral: Reaching Movements
- Reaching Task (Active Comparator): Age-match control participants will make decision while moving
  Interventions: Behavioral: Reaching Movements

INTERVENTIONS:
Behavioral: Reaching Movements — participants will perform a perceptual decision making task while moving their hand.

SUMMARY:
The investigators aim to understand the interplay and neural structures involved with decision--making and movement for participants with mild cognitive impairment. Rapidly deciding and acting becomes bottlenecked with mild cognitive impairment and Alzheimer's, leading to detrimental outcomes such as falling and car crashes. The investigators work will have a tangible impact by discovering sensitive biomarkers to detect disease onset and pave the way for informed and effective neurorehabilitation.

DETAILED DESCRIPTION:
Mild cognitive impairment leads not only to impaired decision making, but also movement deficits that predict the development of Alzheimer's disease. Recent behavioral work has suggested a common mechanism that throttles the speed of both decisions and reaching movements, which is supported by converging neural evidence that finds an interac-tion between decision making and movement (motor) circuits. Yet it remains unknown how the interplay between decision making and motor neural circuits becomes impaired and impedes rapid responses for those with mild cognitive impairment. Here the investigators test the central hypothesis that there is an impaired interaction between decision making and motor neural circuits with mild cognitive impairment.

First, the investigators will use human reaching experiments to establish that mild cognitive impairment disrupts the interplay of decision making and motor control. Second, the investigators will use Magnetic resonance elastography to elucidate whether brain stiffness in decision making and motor brain regions are related to altered movement behavior. The expected outcome is a mechanistic understanding of how impaired decision making and motor neural circuits impact movement for those with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. age 45 - 90 years
2. Perfect or corrected vision
3. Ability to reach
4. Neurotypical Age-Matched control participants - No history of neurological disorders or injury.
5. Mild Cognitive Impairment participants - clinical diagnosis of amnestic mild cognitive impairment.

Exclusion Criteria:

1. Any injury or condition that impacts reaching
2. Traumatic brain injury, such as concussion, in the last 6 months.
3. Neurotypical Age-Matched control participants: Modified Telephone Interview for Cognitive Status (TICS-m) score < 34
4. Mild Cognitive Impairment participants: Modified Telephone Interview for Cognitive Status (TICS-m) score > 34
5. Mild Cognitive Impairment participants: Mini-Mental State Examination Second Edition (MMSE-2) score < 21.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reaching Movements | through study completion, an average of 1 year
  Hand position will be recorded throughout each trial during the behavioral task
Change in brain mechanical properties | through study completion, an average of 1 year
  Investigators are assessing change in brain structure through mechanical properties

SECONDARY OUTCOMES:
Decision Time | through study completion, an average of 1 year
  Decision time will be calculated on each trial during the behavioral task

CONTACTS AND LOCATIONS:
Overall Officials: Josh Cashaback, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No